CLINICAL TRIAL: NCT07020624
Title: Comparison of the Analgesic Effects of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) and Serratus Anterior Plane Block (SAPB) on Postoperative Analgesia in Video-Assisted Thoracoscopic Surgery (VATS)
Brief Title: Serratus Posterior Superior Intekcostal Plane Block vs Serratus Anterior Plane Block for Postoperative Analgesia in VATS: A Randomized Trial"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SPSIPB
Record Dates: First submitted 2025-05-22; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Video Assisted Thoracoscopic Surgery; Postoperative Analgesia
Keywords: serratus posterior superior intercostal plane block; Video-assisted thoracoscopic surgery; serratus anterior plane block

STUDY DESIGN:
Intervention Model Description: two interventional group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The anesthetist who will perform the blocks will not participate in the pain follow-up of the patients. Postoperative pain assessment and data collection will be performed by another anesthetist blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group serratus anterior plane block (SAP) (Active Comparator): At the end of the surgery, ultrasound-guided serratus anterior plane block is performed with 0.25% bupivacaine. Perioperative and postoperative routine analgesic protocol is applied (consisting of intravenous analgesics and intravenous patient-controlled analgesia) without additional intervention (block) Standard Pain Monitoring and Follow-up is performed
  Interventions: Other: SAPB
- group serratus posterior superior intercostal plane block(SPSIP) (Active Comparator): At the end of the surgery, ultrasound-guided serratus posterior superior intercostal plane block is performed with 0.25% bupivacaine. Perioperative and postoperative routine analgesic protocol is applied (consisting of intravenous analgesics and intravenous patient-controlled analgesia) without additional intervention (block) Standard Pain Monitoring and Follow-up is performed
  Interventions: Other: SPSIPB

INTERVENTIONS:
Other: SAPB — Ultrasound guided serratus anterior plane block will be performed.
  Arms: group serratus anterior plane block (SAP)
Other: SPSIPB — Ultrasound guided serratus posterior superior intercostal plane block will be performed.
  Arms: group serratus posterior superior intercostal plane block(SPSIP)

SUMMARY:
Thoracotomy is known as one of the most painful surgical procedures, with up to 65% of patients developing chronic post-thoracotomy pain syndrome (PTPS), and approximately 10% experiencing pain that significantly impacts quality of life. Video-assisted thoracoscopic surgery (VATS) has become increasingly common over the past decade and offers reduced postoperative pain, morbidity, and length of hospital stay compared to open thoracotomy. However, VATS can still cause moderate to severe postoperative pain and a high risk of chronic pain. Optimizing analgesia after VATS remains critical. With advances in ultrasound technology, several regional anesthesia techniques such as serratus anterior plane block (SAPB), erector spinae plane block (ESPB), and thoracic epidural analgesia (TEA) have shown comparable efficacy. In 2023, Tulgar et al. described the serratus posterior superior intercostal plane block (SPSIPB), which demonstrated dermatomal coverage from C3 to T10. This randomized controlled trial aims to compare the analgesic efficacy of SPSIPB and SAPB in patients undergoing VATS procedures.

DETAILED DESCRIPTION:
The patients will be divided into two groups and all will receive general anesthesia. Before extubation, one group will receive a Serratus Anterior Plane Block, and the other group will receive a Serratus Posterior Superior Intercostal Plane Block. The randomization of the study will be performed by a physician who will not be involved in the patient follow-up, using a computer-generated randomization code (generated by the computer). The interfascial plane block (Serratus Anterior Plane Block or Serratus Posterior Superior Intercostal Plane Block) will be given to the anesthesiologist in a sealed envelope by an independent assistant personnel outside the study. The patient will not be aware of which block is being applied. The anesthesiologist performing the block will not participate in the patients' pain monitoring. Postoperative pain assessment and data collection will be performed by another anesthesiologist who is unaware of the study.

For standardization purposes, the block procedure will be performed by an experienced anesthesiologist who has performed at least 20 successful and uncomplicated procedures before.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 35 kg/m² Patients with ASA scores I, II, III

Exclusion Criteria:

* Patients who do not want to be included in the study Psychiatric and neurological disease with blurred consciousness Patients with ASA > 3 BMI > 35 kg/m² Abnormality in coagulation parameters History of allergy to local anesthetic drugs Infection at the injection site Patients whose surgical procedure time exceeds 150 minutes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption in the first 24 hours postoperatively | up to 24 hours
  Morfin consumption in the first 24 hours after surgery

SECONDARY OUTCOMES:
Pain density | up to 24 hours.
  NRS scores (Numeric rating scale; 0: no pain, 10: severe pain) in the first 24 hours after surgery
Quality of recovery | 24 hours after surgery
  QR15 scores
Nausea and vomiting | up to 24 hours
  Nausea and vomiting scores in the first 24 hours (verbal rating scale; 0= none, 1= nausea, 2= gagging, 3= vomiting)
shoulder pain | up to 24 hours
  postoperative shoulder pain;shoulder pain will be evaluated as present/absent

CONTACTS AND LOCATIONS:
Overall Officials: hamiyet şenol çakmak, specialist, Principal Investigator — samsun university Samsun Training and Research Hospital
Locations (1):
- Samsun University,, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No